CLINICAL TRIAL: NCT01875081
Title: Randomized Exploratory Clinical Trial to Evaluate the Safety and Effectiveness of Stem Cell Product in Alcoholic Liver Cirrhosis Patient.
Brief Title: REVIVE(Randomized Exploratory Clinical Trial to Evaluate the Safety and Effectiveness of Stem Cell Product in Alcoholic Liver Cirrhosis Patient)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmicell Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PMC-BD-CT-P-002; NCT01875211 (obsolete NCT alias)
Record Dates: First submitted 2013-06-07; First posted 2013-06-11 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Alcoholic Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis, Alcoholic

ARMS (3):
- Control group (No Intervention): Best Supportive care
- 1-time injection group: Livercellgram (Experimental): Within 1 month after extracting bone marrow, directly inject 5X107 autologous bone marrow-derived mesenchymal stem cells within liver through the hepatic artery.
  Interventions: Biological: Livercellgram
- 2-time injection group: Livercellgram (Experimental): Within 1 month after extracting bone marrow, directly inject 5X107 autologous bone marrow-derived mesenchymal stem cells within liver through the hepatic artery. Within 1 month after cell injection, re-inject autologous bone marrow-derived mesenchymal stem cells.
  Interventions: Biological: Livercellgram

INTERVENTIONS:
Biological: Livercellgram — Livercellgram
  * Dosage form and appearance: White cell suspension is filled in a clear plastic syringe, and fixed with an occlude on the prefilled syringe tip ② Component: Autologous bone marrow-derived mesenchymal stem cell ③ Amount: 5X107 cells, 1-time or 2-time injection ④ Storage Method: Stored in airtight container at 20~25℃
    * Injection Method: Directly inject into liver through hepatic artery
  Other Names: Autologous bone marrow-derived mesenchymal stem cell
  Arms: 1-time injection group: Livercellgram; 2-time injection group: Livercellgram

SUMMARY:
If the participant voluntarily agrees to participate in the clinical trial before registration, the investigator conducts a screening test to evaluate the participant's suitability.

A participant that satisfies all selection and exclusion criteria is assigned randomly to a test group (1-time or 2-time injection group) or control group (no-cell therapy group). Participants assigned to the 1-time injection group conduct cell therapy within 1 month after bone marrow aspiration. Before implementing cell therapy, implement hepatic artery catheterization which inserts a catheter into the hepatic artery through the right aorta femoralis and inject 5X107 autologous bone marrow-derived mesenchymal stem cells. Participants assigned to the 2-time injection group store 1-time injection amount of mesenchymal stem cells while being cultivated after sampled from the bone marrow, and will re-inject autologous mesenchymal stem cells within 1 month after first injection.

Participants will make a total of 8 hospital visits on a 4-week interval after registration, and effectiveness and safety will be evaluated based on a fixed procedure on every visit.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or clinically diagnosed as alcoholic liver cirrhosis
2. Classified as Child-Pugh grade B or C
3. Age of 20 ~ 70 years
4. Capable of conducting hepatic artery catheterization which inserts a catheter up to the hepatic artery
5. In the case of fertile women, confirmed as negative in pregnancy test when screening, and agreed to avoid pregnancy during the trial period
6. Women capable of pregnancy must satisfy the following conditions; Has been through menopause for at least 1 year, has no possibility of pregnancy via surgery/procedure, or effectively used acceptable contraceptive methods (Intrauterine device-loop, mirena, diaphragm or condom/femidom, oral contraceptive pills, non-oral contraceptives)
7. Patient who can agree to participate in the clinical trial by oneself or by one's legal representative
8. Able to conduct the clinical trial according to the protocol

Exclusion Criteria:

1. Diagnosed with malignant hematologic disease (acute myeloid leukemia, acute lymphoblastic leukemia, non-Hodgkin lymphoma, Hodgkin lymphoma, multiple myeloma) and not cured from it
2. Patient with severe aplastic anemia
3. Has a medical record of solid cancer(within 5 years prior to screening), or diagnosed with solid cancer and currently receiving cancer treatment
4. Incapable of conducting hepatic artery
5. Patient who consumed alcohol and took hepatotoxic drugs within 6 months prior to registration
6. Has continuously taken a large amount of steroids or antibiotics for 1 month prior to registration
7. Judged by a researcher to have had major orthopedic surgery, organ biopsy, or similar external injury within 3 months prior to registration
8. Evidence of active autoimmune liver disease
9. Patient with extrahepatic biliary stricture
10. Patient who conducted transjugular intrahepatic portosystemic shunt
11. Has active thrombosis of the portal or hepatic veins
12. Patient with sepsis
13. Patient who suffers heart, renal, respiratory failure
14. Patient who is positive in pathogenic test (HIV, Syphilis,HBV,HCV)
15. Pregnant or lactating woman
16. Patient who cannot adapt to the protocol and follow-up observation
17. Patient who has experienced drug abuse for the past 1 year
18. Participated in the other clinical trials within 30 days before registration
19. Patient with any disease or condition which the investigator feel would interfere with trial or the safety of the subject

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Histopathological evaluation (Fibrosis Grade - Laennec Scoring System) | 6 month after cell therapy

SECONDARY OUTCOMES:
Histopathological evaluation score (Ratio of 1-time injection group to 2-time injection group comparison) | 6month
MELD Score | 6month
Child-Pugh grade | 6month
Liver Function Test (ALT, AST, ALP, Albumin, billirubin, r-GT) | 6month
Visual Inspection (Liver volume, Fibroscan) | 6month

CONTACTS AND LOCATIONS:
Overall Officials: Soon Koo Baik, M.D.,Ph.D, Principal Investigator — Yonsei University, Wonju Christian Hospital; Si-Hyun Bae, M.D.,Ph.D, Principal Investigator — The Catholic University of Korea
Locations (1):
- Pharmicell Co., Ltd., Seoul, South Korea